CLINICAL TRIAL: NCT05500391
Title: Randomized Phase II Trial Evaluating Compliance With Monitoring Conducted Either by a Hospital-based Physician in Person or by a Nurse in Remote Monitoring
Brief Title: Assessment of Compliance With Monitoring Conducted by a Physician in Person or by a Nurse in Remote Monitoring
Acronym: SUR-CAN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Canceropôle Nord Ouest (Other); Groupement Interrégional de Recherche Clinique et d'Innovation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SUR-CAN-2201
Record Dates: First submitted 2022-08-10; First posted 2022-08-15 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Stage I Testicular Seminoma; Stage I Testicular Nonseminomatous Germ Cell Tumor; Gastrointestinal Stromal Tumors; Ovarian Germ Cell Tumor; Adenocarcinoma, Clear Cell; Borderline Ovarian Tumor; Sex Cord-Stromal Tumor; Mucinous Adenocarcinoma of Ovary; Carcinoma, Small Cell; Carcinosarcoma, Ovarian; Serous Tumor of Ovary; Glioma; Neuroendocrine Tumors; Aggressive Fibromatosis of Abdominal Wall (Disorder)
MeSH Terms: conditions — Seminoma; Gastrointestinal Stromal Tumors; Adenocarcinoma, Clear Cell; Sex Cord-Gonadal Stromal Tumors; Carcinoma, Small Cell; Carcinosarcoma; Glioma; Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Telesurveillance by a nurse
  Interventions: Other: Oncological Follow-up
- Control (Other): On-site surveillance by a hospital physician
  Interventions: Other: Oncological Follow-up

INTERVENTIONS:
Other: Oncological Follow-up — Post-cancer surveillance (including biological, clinical and imaging exams depending on the condition)

SUMMARY:
This is a multicenter, interventional, randomized study among adult patients recently diagnosed with a rare tumor (<12 months). The study will aim to compare compliance with the personalized post-treatment surveillance plan, established for each patient according to national guidelines, when the surveillance is conducted in person by a hospital-based physician (control arm) or remotely by a trained nurse (experimental arm).

DETAILED DESCRIPTION:
The primary objective of this study is to compare 2-year compliance with the personalized post-treatment surveillance plan between the two arms.

The secondary objectives are to compare between the two arms :

* Long-term compliance (5-year follow-up)
* Use of care
* Oncological events and their management
* Supportive care needs

The exploratory objectives are to :

* Evaluate the costs in terms of medical transportation
* Evaluate and compare patients' satisfaction and psychological well-being (in terms of anxiety/depression)
* Evaluate the homogeneity of the impact of the intervention according to covariates (gender, tumor pathology, occupational status, and center)
* Evaluate the reasons for recruitment failures

ELIGIBILITY:
Inclusion Criteria:

* Positive diagnosis (anatomopathology) of tumor within 12 months
* Patient 18 years of age or older
* Patient with one of the following conditions:

  1. Desmoid fibromatosis of the abdominal wall operated on or under active surveillance
  2. Stage I testicular seminoma (whether or not treated with carboplatin AUC7)
  3. Stage I non-seminomatous germ cell tumor (with or without adjuvant BEP chemotherapy)
  4. Operated GIST with low risk of relapse
  5. Rare gynecological tumors (sex cord and stromal tumors; germ cell tumors of the ovary, clear cell adenocarcinoma, mucinous adenocarcinoma of the ovary, borderline tumors, small cell carcinoma, ovarian and uterine carcinosarcoma, low grade serous tumors), operated
  6. Low-grade glioma, operated
  7. Low-grade neuroendocrine tumor, treated by surgery alone
* Patient who has given consent to participate in the study

Exclusion Criteria:

* Contraindication to imaging tests required for the surveillance plan
* No telephone
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
2-year compliance to the customized surveillance plan | 2 years
  Compliance is defined by completion of all scheduled examinations (telephone contact, biological, clinical examination and imaging examination) with a margin of + or - 30 days from the scheduled date

SECONDARY OUTCOMES:
5-year compliance to the customized surveillance plan | 5 years
  Compliance is defined by completion of all scheduled examinations (telephone contact, biological, clinical examination and imaging examination) with a margin of + or - 30 days from the scheduled date
Drop-out rate | 5 years
  Rate of patients lost to follow-up or quitting the surveillance program
Description of the use of care | 5 years
  * number of physical consultations at the investigator site
  * number of emergency room visits for oncological reasons
  * number of extra-hospital consultations for oncological reasons
Occurrence and management of oncological events | 5 years
  Occurence and type of oncological event : relapse/progression.
  The management of oncological events will be evaluated according to three criteria :
  * completion of an oncological surgery
  * implementation of a treatment by radiotherapy
  * implementation of a systemic therapy such as chemotherapy
Progression-free survival | 5 years
  Time from randomization to first oncological event (progression/relapse) or death from any cause.
Overall survival | 5 years
  Time from randomization to death from any cause
Support care needs identified | 2 years (early termination in case of relapse of the disease)
  Support care needs include :
  * algology consultation
  * nutrition/diet consultation
  * psycho-oncology consultation
  * social worker consultation
  * job retention consultation

OTHER OUTCOMES:
Costs in terms of medical transport use | 5 years
  Medical transport includes light medical vehicles and ambulances
Salary mass mobilized from a hospital perspective in both arms | 5 years
  Salary mass mobilized from a hospital perspective in both arms
Patient satisfaction | 2 years
  Patients will answer a satisfaction survey (French Version of the Princess Margaret Hospital Satisfaction With Doctor) at different points of the study depending on their pathology
Patient reported outcomes | 2 years
  Patient reported outcomes will be evaluated using the Hospital Anxiety and Depression Scale (HADS) questionnaire at different points of the study depending on their pathology.
  The questionnaire consists of a list of questions to determine the level of anxiety and depression experienced by the patients. Each question is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression:
  A score equal to or less than 7 indicates no symptoms, A score of 8 - 10 indicates a questionable symptoms, A score of 11 and above confirms of the presence of anxiety and/or depression symptoms.
Evaluation of the causes of recruitment failures | During the recruiting period (18 months)
  In each investigating site, a screening log will be completed to find out the reasons for recruitment failures

CONTACTS AND LOCATIONS:
Overall Officials: PENEL Nicolas, MD, PhD, Principal Investigator — Centre Oscar Lambret
Locations (3):
- France (3):
  - CHU Amiens, Amiens
  - Centre François Baclesse, Caen
  - Centre Oscar Lambret, Lille

REFERENCES:
- [Background] Kimman ML, Bloebaum MM, Dirksen CD, Houben RM, Lambin P, Boersma LJ. Patient satisfaction with nurse-led telephone follow-up after curative treatment for breast cancer. BMC Cancer. 2010 Apr 30;10:174. doi: 10.1186/1471-2407-10-174. PMID 20429948
- [Background] Moloney J, Partridge C, Delanty S, Lloyd D, Nguyen MH. High efficacy and patient satisfaction with a nurse-led colorectal cancer surveillance programme with 10-year follow-up. ANZ J Surg. 2019 Oct;89(10):1286-1290. doi: 10.1111/ans.15333. Epub 2019 Jul 7. PMID 31280494
- [Background] Martin E, Persaud S, Corr J, Casey R, Pillai R. Nurse-led active surveillance for prostate cancer is safe, effective and associated with high rates of patient satisfaction-results of an audit in the East of England. Ecancermedicalscience. 2018 Jul 25;12:854. doi: 10.3332/ecancer.2018.854. eCollection 2018. PMID 30093916
- [Background] Keshava HB, Tan KS, Dycoco J, Huang J, Berkowitz A, Sumner D, Devigne A, Adusumilli P, Bains M, Bott M, Isbell J, Downey R, Molena D, Park B, Rocco G, Sihag S, Jones DR, Rusch VW. Long-term assessment of efficacy with a novel Thoracic Survivorship Program for patients with lung cancer. J Thorac Cardiovasc Surg. 2022 May;163(5):1645-1653.e4. doi: 10.1016/j.jtcvs.2021.11.026. Epub 2021 Nov 20. PMID 34922758
- [Background] Ferrua M, Minvielle E, Fourcade A, Lalloue B, Sicotte C, Di Palma M, Mir O. How to Design a Remote Patient Monitoring System? A French Case Study. BMC Health Serv Res. 2020 May 19;20(1):434. doi: 10.1186/s12913-020-05293-4. PMID 32429987